CLINICAL TRIAL: NCT02553044
Title: Change in Free 25(OH)D After High Dose in Vitamin D Deficient Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: National Osteoporosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STH18850
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Vitamin D Deficiency; Osteoporosis
MeSH Terms: conditions — Vitamin D Deficiency; Osteoporosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 50 000IU Vitamin D3 (Experimental): 50 000IU oral vitamin D3 (cholecalciferol) administered at baseline only.
  Interventions: Dietary Supplement: Cholecalciferol (Vitamin D3)
- 150 000IU Vitamin D3 (Experimental): 150 000IU oral vitamin D3 (cholecalciferol) administered at baseline only.
  Interventions: Dietary Supplement: Cholecalciferol (Vitamin D3)
- 500 000IU Vitamin D3 (Experimental): 500 000IU oral vitamin D3 (cholecalciferol) administered at baseline only.
  Interventions: Dietary Supplement: Cholecalciferol (Vitamin D3)
- Concurrent Control (No Intervention): Control group to receive no intervention.

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (Vitamin D3) — Oral vitamin D3 doses made up using 50 000IU ampules of vitamin D3 dissolved in 1ml of olive oil.
  Other Names: Invita D3
  Arms: 150 000IU Vitamin D3; 50 000IU Vitamin D3; 500 000IU Vitamin D3

SUMMARY:
Total 25(OH)D is currently used as a biomarker of vitamin D status. However, there is some debate as to whether total 25(OH)D is the best marker to use.

It has been suggested that free vitamin D may be better because it may be more biologically available.

There are also some uncertainties about how we treat vitamin D deficiency. A single dose is attractive because it is certain that the patient has had the dose and there is no requirement for ongoing compliance, but it is still not clear what the best dose is to give. Also, recent studies have highlighted that high dose vitamin D supplementation may increase the risk of falling in older populations.

The investigators believe that studying how free vitamin D responds to different bolus doses is the best way address some of the current research gaps, including what is the best biomarker of vitamin D status, what is the mechanism of vitamin D toxicity and what is a safe bolus dose to treat deficiency.

The investigators will study changes in total and free 25(OH)D, and also clinical response, to three different bolus doses of vitamin D (50 000IU, 150 000IU and 500 000IU) in 84 vitamin D deficient postmenopausal women, over a three month period with 5 study visits. A concurrent control group of 28 vitamin D sufficient postmenopausal women will also be recruited.

This will allow the investigators to determine how total and free vitamin D change with bolus dosing and whether there is a disproportionate rise in free 25(OH)D with higher doses that may lead to hypercalcemia and falls.

DETAILED DESCRIPTION:
The most commonly used measurement of vitamin D status is serum 25-hydroxyvitamin D (25(OH)D). However there is no clear consensus on the level of 25(OH)D required to protect against adverse effects of deficiency.

One approach is to define deficiency is the level of 25(OH)D at which there is a secondary physiological response, such as a rise in parathyroid hormone. However, this approach has not yielded a clear answer. Total 25(OH)D below 30nmol/l is not always associated with an increased parathyroid hormone (PTH) response, and total 25(OH)D and PTH do not always respond to vitamin D supplementation. This suggests that total 25(OH)D measurement may not be the best biological marker of vitamin D status.

Vitamin D and its metabolites are bound to proteins in the circulation: around 85-90% of 25(OH)D is bound to vitamin D binding protein (DBP), 10-15% is bound to albumin, and less than 1% is in the free form. DBP protects 25(OH)D from degradation and allows a circulating store to accumulate.

The free hormone hypothesis suggests that only the unbound 'free' portion of protein bound hormones is biologically active, and that this should be measured for the accurate assessment of hormone availability. Calculated free 25(OH)D concentrations have been shown to be better correlated to bone mineral density (BMD) than total 25(OH)D in a healthy population and to be more closely related to PTH in patients with end stage renal disease.

The binding capacity of DBP may be overwhelmed in some situations. In female participants treated with an oral dose of 500,000 IU annually for 3 years there was an increase in the risk of falls and fractures that was particularly marked in the three month period after each dose. It has been proposed that there was vitamin D toxicity and possible hypercalcaemia during this period due to the binding capacity of DBP being overwhelmed by the large increase in 25(OH)D with a relatively greater increase in free 25(OH)D. However, free vitamin D and calcium were not measured in the study, so there is not yet evidence to support this hypothesis.

The investigators will study changes in total and free 25(OH)D, and clinical response to three different bolus doses of vitamin D (50,000 units, 150,000 units and 500,000 units) in 84 vitamin D deficient (<30nmol/l) postmenopausal women over three months. This will allow the investigators to determine how free and total 25(OH)D change with bolus dosing and whether there is a disproportionately high rise in free 25(OH)D with higher doses. This will also generate a better understanding of what the optimum bolus dose for treatment of vitamin D deficiency is and whether free 25(OH)D may be a better marker of vitamin D status in some situations.

Aims of the study:

* To determine the effect of three different vitamin D bolus doses on free 25(OH)D and total 25(OH)D in vitamin D deficient post-menopausal women.
* To determine the effect of different vitamin D bolus doses on parameters of calcium metabolism, bone turnover markers and physical function in vitamin D deficient post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* 25(OH)D < 30nmol/l for treatment groups or 25(OH)D >50nmol/l for control group
* BMI between 20 kg/m2 and 30kg/m2
* 55 years and over and postmenopausal (at least 5 years since last menstrual period)
* Able and willing to participate in the study and provide written informed consent.

Exclusion Criteria:

* History of any long term immobilization (duration greater than three months)
* Pre-diagnosed diabetes mellitus
* High trauma fracture or low trauma fracture less than one year prior to recruitment
* History of or current conditions known to affect vitamin D or bone metabolism, including:

Chronic renal disease Malabsorption syndromes Diagnosed endocrine disorders Hypercalcaemia Diagnosed restrictive eating disorder

* Use of medications or treatment known to affect vitamin D or bone metabolism such as bisphosphonates or anti-epileptic medication.
* Alcohol intake of greater than 21 units per week
* Holiday with significant sunlight exposure in the last six weeks
* Planned sun holiday within study period
* Abnormal clinical laboratory parameters that are assessed as clinically significant by the PI.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Free 25(OH)D | Baseline to visit 3 (5-7 days after administration)
  Change in free 25(OH)D from baseline to visit 3 (5-7 days after administration)

SECONDARY OUTCOMES:
Proportion of total 25(OH)D to free 25(OH)D | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between-group difference in proportion of serum free 25(OH)D to total 25(OH)D at 5, 28 days and 84 days
1, 25(OH)2D | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between-group difference in 1, 25(OH)2D at 5, 28 days and 84 days
Ionized calcium | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between-group difference in ionized calcium at 5, 28 days and 84 days
Parathyroid Hormone | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between-group difference in PTH at 5, 28 days and 84 days
Bone turnover marker - Alkaline Phosphatase | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between group difference in alkaline phosphatase at 5, 28 and 84 days
Bone turnover marker - CTX | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between group difference in CTX at 5, 28 and 84 days
Bone turnover marker - PINP | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between group difference in PINP at 5, 28 and 84 days
Bone turnover marker - Osteocalcin | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between group difference in Osteocalcin at 5, 28 and 84 days
Repeated chair stand test score | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between group difference in repeated chair stand test score at 5, 28 and 84 days
Tandem stand balance test score | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between group difference in tandem stand balance test score at 5, 28 and 84 days
8-feet walk course test score | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between group difference in 8-feet walk course test score at 5, 28 and 84 days
Laying blood pressure | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between group difference in laying blood pressure at 5, 28 and 84 days
Standing blood pressure | 5(+/-2) days, 28(+/-3) days and 84(+/-5) days
  Between group difference in standing blood pressure at 5, 28 and 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Walsh, MBChB, PhD, Principal Investigator — University of Sheffield
Locations (1):
- Clinical Research Facility, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Background] Shibli-Rahhal A, Paturi B. Variations in parathyroid hormone concentration in patients with low 25 hydroxyvitamin D. Osteoporos Int. 2014 Jul;25(7):1931-6. doi: 10.1007/s00198-014-2687-4. Epub 2014 Mar 20. PMID 24647889
- [Background] Sanders KM, Stuart AL, Williamson EJ, Simpson JA, Kotowicz MA, Young D, Nicholson GC. Annual high-dose oral vitamin D and falls and fractures in older women: a randomized controlled trial. JAMA. 2010 May 12;303(18):1815-22. doi: 10.1001/jama.2010.594. PMID 20460620
- [Background] Powe CE, Ricciardi C, Berg AH, Erdenesanaa D, Collerone G, Ankers E, Wenger J, Karumanchi SA, Thadhani R, Bhan I. Vitamin D-binding protein modifies the vitamin D-bone mineral density relationship. J Bone Miner Res. 2011 Jul;26(7):1609-16. doi: 10.1002/jbmr.387. PMID 21416506
- [Background] Bhan I, Powe CE, Berg AH, Ankers E, Wenger JB, Karumanchi SA, Thadhani RI. Bioavailable vitamin D is more tightly linked to mineral metabolism than total vitamin D in incident hemodialysis patients. Kidney Int. 2012 Jul;82(1):84-9. doi: 10.1038/ki.2012.19. Epub 2012 Mar 7. PMID 22398410